CLINICAL TRIAL: NCT03242408
Title: Dosing Flexibility Study of Oral Testosterone Undecanoate (TU, LPCN 1021) in Hypogonadal Men.
Brief Title: Dosing Flexibility Study of Oral Testosterone Undecanoate (TU, LPCN 1021)
Acronym: DF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lipocine Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPCN 1021-16-003
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Results first posted 2019-09-11 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-08

CONDITIONS: Hypogonadism, Male
MeSH Terms: conditions — Eunuchism | interventions — Testosterone Propionate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral testosterone undecanoate, LPCN 1021 (Experimental): Oral testosterone undecanoate, LPCN 1021 150 mg TU three times a day
  Interventions: Drug: LPCN 1021

INTERVENTIONS:
Drug: LPCN 1021 — Oral testosterone undecanoate

SUMMARY:
This is a multicenter, open-label, one treatment study evaluating the efficacy of LPCN 1021 in adult hypogonadal male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Serum total T below 300 ng/dL based on 2 consecutive blood samples obtained between 6 and 10 AM, on two separate days at approximately the same time of day, following an appropriate washout of current androgen replacement therapy.
2. Subjects should be diagnosed to be primary (congenital or acquired) or secondary hypogonadal (congenital or acquired).
3. Naïve to androgen replacement or has discontinued current treatment and completed adequate washout of prior androgen therapy. Washout must be completed prior to collection of baseline serum T samples to determine study eligibility.

Exclusion Criteria:

1. History of significant sensitivity or allergy to androgens, or product excipients.
2. Clinically significant findings in the pre-study examinations including abnormal breast examination requiring follow-up.
3. Abnormal prostate digital rectal examination (DRE) with palpable nodule(s).
4. Subjects with symptoms of moderate to severe benign prostatic hyperplasia.
5. Clinically significant abnormal laboratory value, in the opinion of the investigator, in serum chemistry, hematology, or urinalysis
6. Positive test result for hepatitis A virus immunoglobulin M (HAV-IgM), hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus antibodies (HIV Ab).
7. History of gastric surgery, cholecystectomy, vagotomy, bowel resection or any surgical procedure that might interfere with gastrointestinal motility, pH or absorption.
8. History of any clinically significant illness, infection, or surgical procedure within 1 month prior to study drug administration.
9. History of stroke or myocardial infarction within the past 5 years.
10. History of or current or suspected prostate or breast cancer.
11. History of untreated and severe obstructive sleep apnea.
12. History of long QT syndrome (QTc > 450) or unexplained sudden death in a first degree relative (parent, sibling, or child).

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony DelConte, MD, Study Director — Lipocine Inc.

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Testosterone Undecanoate, LPCN 1021
Started | 100
Completed | 98
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Oral Testosterone Undecanoate, LPCN 1021
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 91
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 100
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 84
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 100
Baseline Testosterone Value (ng/dL) [Mean (Standard Deviation); unit: ng/dL] | 189 (72.4)

OUTCOME MEASURES:

1. Primary Outcome: Percent of LPCN 1021-treated Subjects Who Achieve a Total Testosterone Average Concentration [Cavg] in the Normal Range
Description: Safety Set; Proportion of LPCN 1021-treated subjects who achieve a total testosterone average concentration [Cavg] in the normal range
Time Frame: Following 24 days of treatment
Population: Safety Set
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Oral Testosterone Undecanoate, LPCN 1021
Number analyzed (Participants) | 100
Percent of participants | 69 [60 to 78]

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Oral Testosterone Undecanoate, LPCN 1021
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 9/100
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Testosterone Undecanoate, LPCN 1021 (N=100)
Edema Peripheral (Metabolism and nutrition disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hyperhidrosis (Nervous system disorders) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Tooth Fracture (Gastrointestinal disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Hypertension (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT03242408/Prot_SAP_000.pdf